CLINICAL TRIAL: NCT04465409
Title: Evaluation of Safety and Efficacy of Intrastromal Implantation of CorVision® Bioengineered Corneal Inlay for Correction of Presbyopia.
Acronym: CorVision
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LinkoCare Life Sciences AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG-PRT-002-Rev6
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Presbyopia
Keywords: presbyopia; bioengineered corneal inlay; femto second laser; intrastromal implantation; biocompatible; medical device; sterile; medical grade; natural; refractive error
MeSH Terms: conditions — Presbyopia; Infertility; Refractive Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Presbyopic adults (Experimental): Presbyopic adults, male or female between 40-65 years of age who need from +1.25 D to +3.50 D of reading addition in the non-dominant eye to improve near visual acuity by at least one line or more.
  In this investigation, CorVision® will be implanted in the non-dominant eye to improve near vision and the dominant eye is left intact or corrected by a standard refractive surgery to emmetropia. In brief, subjects will undergo laser corneal surgery on their non-dominant eye to create an anterior stromal pocket into which the investigational device will be implanted.
  Interventions: Device: Intrastromal implantation of CorVision bioengineered corneal inlay for correction of presbyopia.

INTERVENTIONS:
Device: Intrastromal implantation of CorVision bioengineered corneal inlay for correction of presbyopia. — Presbyopia is an age-related progressive loss of crystalline lens accommodation power resulting in the decreased ability to see near objects. CorVision® is a tissue-mimetic device primarily intended to be used as a corneal inlay in the management of presbyopia and low hypermetropia. The inlay is inserted into the patient's cornea via a minimally invasive laser pocket procedure to modify corneal surface topography and corneal optical performance.

SUMMARY:
This clinical investigation is a prospective, multicentre, non-comparative case series to assess safety and efficacy of CorVision® bioengineered corneal inlay for improving uncorrected near vision in presbyopic subjects.

In this study a sterile medical grade collagen-based bioengineered corneal inlay (CorVision®), which closely mimics the human corneal tissue, will be tested as a natural microlens for correction of near vision in presbyopic patients. The primary endpoint for this study is to further determine the safety of the inlay and the secondary endpoint is to determine the efficacy of the inlay to improve uncorrected near vision.

CorVision® implantation will be done via a minimally invasive laser-assisted intra-stromal surgery. Besides important information concerning details of the surgical method and postoperative care, tolerance of the device and possible adverse events will be reported along with several clinical parameters to be measured preoperatively and postoperatively. The study will consist of 110 subjects receiving the inlay to be included within a recruitment period of 18 months at multiple clinical sites. All subjects will be followed for minimum 12-months postoperatively. Postoperative evaluations are scheduled at 1 week, 1, 3, 6, and 12 months.

DETAILED DESCRIPTION:
Upon signing of informed consent and study inclusion, both eyes will be screened to determine which eye is dominant and to ensure that the non-dominant eye meets the visual acuity, refraction, and other inclusion criteria. In this investigation, the monovision concept will be utilized, e.g. CorVision® will be implanted in the non-dominant eye to improve near vision and the dominant eye is left intact or corrected by a standard refractive surgery to emmetropia. In brief, subjects will undergo laser corneal surgery on their non-dominant eye to create an anterior stromal pocket into which the investigational device will be implanted. Combined antibiotic - steroid eye drops will be instilled for 4 weeks post-implantation.

The investigational treatment does not introduce foreign cells into the patient, requires only a short course of local immunosuppression (4 weeks compared to 12 months or longer for some other treatment options), and is reversible as the investigational device can be removed later if required. Moreover, should serious intra-operative or post-operative complications arise during or following implantation of the investigational device that cannot be treated with medications (for example thinning or clouding of the cornea), the CorVision® device can be removed and the patient can undergo standard-of-care for complications after laser surgery.

Following implantation of the CorVision®, postoperative eye examinations will be conducted at 1 week, 1 month, then at month 3, 6, and 12 and outside of these standard examination times on an as-needed basis at any time. Examinations will include corneal tomography, central corneal thickness, slit lamp corneal transparency, keratometry, anterior segment optical coherence tomography, and general ophthalmic examination including tear break up time, refraction, uncorrected and corrected distance, intermediate and near visual acuity, and in some eyes aberrometer measurements, defocus curve or contrast sensitivity.

The proof-of-concept and feasibility to implant CorVision® by standard surgical methods such as a femto-second assisted pocket surgery and postoperative treatment and assessment protocol for this new medical device have already been developed via prior pre-clinical evaluations and some pilot clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Presbyopic adults, Male or female between 40-65 years of age who need from +1.25 D to +3.50 D of reading addition in the non- dominant eye to improve near visual acuity by at least one line or more.
* Manifest refraction spherical equivalent (MRSE) between -0.75 and +1.50 D with ≤1.5 D of refractive cylinder in the non-dominant eye.
* Stable refraction, i.e. MSRE within 0.50 D over prior 12 months in the non-dominant eye.
* Corrected distance visual acuity CDVA ≥ 0.7 in the dominant and non-dominant eye

Exclusion Criteria:

* Anterior segment pathology in the non-dominant eye.
* Signs or symptoms of clinically significant cataracts in the non-dominant eye.
* Residual, recurrent, active ocular or uncontrolled eyelid disease, or any corneal abnormality (including endothelial dystrophy, recurrent corneal erosion, etc.) in the nondominant eye.
* Visually significant macular pathology
* Central corneal thickness <470 microns in either eye and corneal curvature ≥ 50D
* Corneal ectasia, keratoconus or form frust keratoconus
* Clinically significant dry eye disease
* Any prior ocular surgery in the non-dominant eye.
* History of herpes zoster or herpes simplex keratitis in the non-dominant eye.
* Inability of patient to understand the study procedures and thus inability to give informed consent.
* Participation in another clinical study within the last 3 months
* Already included once in this study (can only be included for one treated eye).
* General history judged by the investigator to be incompatible with the study (e.g., life-
* threatening patient condition, other condition where postoperative follow-up may be difficult).
* known uncontrolled diabetes or other neuro-degenerative disorder (as corneal nerves can be affected leading to impaired wound healing)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2022-09-25 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Safety outcome | 6 months
  The primary safety endpoint is defined such that a rejection leading to implant removal should occur in no more than 3% of implanted eyes. The implant rejection is defined as a clinical situation when the implanted eye has decreased central corneal clarity and decreased implant clarity, corneal vascularization inside of laser created pocket and inflammation.
Efficacy outcome | 6 months
  The primary efficacy endpoint is that more than 65% of the eyes should have an uncorrected near visual acuity (UNVA) of 0.3 logMAR or better at 6 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Katerina Klimesova, MD, Principal Investigator — Gemini Eye Clinics
Locations (1):
- Gemini Eye Clinics, Zlín, Czechia